CLINICAL TRIAL: NCT01871675
Title: An Open-label, Phase Ib Study of IPI-145 in Combination With Rituximab or Bendamustine/Rituximab in Select Subjects With Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: Study of IPI-145 in Combination With Rituximab or Bendamustine/Rituximab in Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI HEMREF 34
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma; Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma; T-cell Lymphoma
Keywords: Lymphoma; Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma; T-cell Lymphoma; Rituxan; Bendamustine; Hematologic Malignancy; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Hematologic Neoplasms; Recurrence | interventions — duvelisib; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: IPI-145 plus Rituximab (Experimental): IPI-145 will be administered orally, twice daily, in 28-day (4-week) cycles, on a continuous basis at the maximum tolerated dose of 25 mg twice-daily (BID), as determined in the dose escalation phase. Twelve (12) cycles of IPI-145 will be administered. Patients who benefit from treatment may continue on study for additional cycles until toxicity or progressive disease.
  Rituximab 375 mg/m2 will be administered intravenously (IV) beginning on Day 1 once weekly during a 28 day cycle; 2 cycles of rituximab will be administered.
  Interventions: Drug: IPI-145; Drug: Rituximab
- Arm 2: IPI-145 plus Rituximab/Bendamustine (Experimental): IPI-145 will be administered orally, twice daily, in 28 day cycles, on a continuous basis, until disease progression, unacceptable toxicity or patient refusal. The maximum tolerated dose of IPI-145 will be 25 mg twice-daily (BID) as determined in the dose escalation phase. Twelve (12) cycles of IPI-145 will be administered. Patients who benefit from treatment may continue on study for additional cycles until toxicity or progressive disease.
  Rituximab 375 mg/m2 will be administered intravenously (IV) beginning on Day 1 once weekly of each 28 day cycle. A maximum of 6 cycles of rituximab will be given. Bendamustine 90 mg/m2 IV will be administered on Days 1 and 2, of each 28 day cycle. Rituximab should be administered prior to bendamustine.
  Interventions: Drug: IPI-145; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: IPI-145
  Other Names: Duvelisib
Drug: Rituximab
  Other Names: Rituxan
Drug: Bendamustine
  Other Names: Treanda
  Arms: Arm 2: IPI-145 plus Rituximab/Bendamustine

SUMMARY:
The goal of this study is to characterize the safety, maximum tolerated dose (MTD) and preliminary efficacy profile of IPI-145 given in combination with rituximab, or bendamustine plus rituximab, to subjects with select relapsed/refractory hematologic malignancies.

DETAILED DESCRIPTION:
This trial consists of two parallel arms. For each treatment arm, a 3+3 dose escalation design will be applied in 3-6 subject cohorts until the maximum tolerated dose of IPI-145 when given with rituximab (Arm 1) or in combination with rituximab and bendamustine (Arm 2) is determined. Treatment arm selection will be chosen by the investigator and will depend on the agents previously administered to the subject. Once the MTD has been determined, the arms will move on to a dose expansion phase. During the dose expansion phase, each treatment arm will enroll to population specific cohorts to assess efficacy. All subjects must have had at least one prior anticancer treatment. The dose expansion cohorts are:

Arm 1: Cohort A - CLL: Cohort B - CD20+ NHL

Arm 2: Cohort A - CLL: Cohort B - CD20+ NHL

ELIGIBILITY:
Inclusion Criteria:

1. Dose Escalation Phase

   Arm 1 and Arm 2: Limited to subjects diagnosed with low grade CD-20 positive B-Cell NHL with at least one prior anticancer treatment.
2. Dose Expansion Phase

   Arm 1 Cohort A: Limited to subjects with CD-20 positive CLL with at least one prior anticancer treatment.

   Arm 1 Cohort B: Limited to subjects with diagnosis of CD-20 positive NHL with at least one prior anticancer treatment.

   Arm 2 Cohort A: Limited to subjects with CD-20 positive CLL with at least one prior anticancer treatment.

   Arm 2 Cohort B: Limited to subjects with diagnosis of CD-20 positive NHL with at least one prior anticancer treatment.
3. Disease status requirement:

   * CLL subjects: symptomatic disease that mandate treatment;
   * Indolent NHL subjects: symptomatic disease requiring treatment according to the clinical judgment of the investigator;
   * Other lymphoma subjects: disease requiring treatment according to the judgment of the investigator.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤2.
5. Subject must have measurable disease using the disease-specific response criteria for NHL or CLL
6. Age ≥ 18 years.
7. Subject has recovered from all clinically significant toxicities related to prior antineoplastic therapies with the exception of alopecia and bone marrow and organ functions.
8. Adequate organ system function ≤2 weeks prior to Day 1, defined as follows:

   * Absolute neutrophil count (ANC) ≥1.0 x 109/L unless related to underlying CLL or indolent NHL bone marrow involvement, and then ANC ≥500 x 109/L permitted.
   * Platelets ≥100 x 109/L unless related to underlying CLL or indolent NHL bone marrow involvement, and then platelets ≥75 x 109/L permitted.
   * Subjects receiving IPI-145 plus rituximab with bone marrow involvement may enroll with platelets ≥40 x 109/L.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 x ULN and total bilirubin ≤1.5 times the upper limit of normal (ULN) (except for subjects with Gilbert's disease)
   * Serum creatinine ≤1.5 x ULN
9. Life expectancy of ≥12 weeks.
10. Women of child-bearing potential (WCBP) must have a negative serum or urine pregnancy test.
11. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Prior allogeneic hematopoietic stem cell transplant (HSCT).
2. Prior autologous transplant or radioimmunotherapy ≤6 months prior to the first dose of trial treatment.
3. Subject has a high grade lymphoma such as Burkitt's, lymphoblastic or small non-cleaved cell lymphomas. Subjects with intermediate grade lymphoma (such as diffuse large B-cell lymphoma) are eligible.
4. Subjects with diffuse B-cell lymphoma must either not be eligible for autologous bone marrow transplant (BMT) or relapsed after autologous BMT.
5. More than three previous cytotoxic chemotherapy regimens for subjects treated on the arm containing bendamustine.
6. Subjects who have had a severe allergic or anaphylactic reaction to any humanized or murine monoclonal antibodies.
7. Chemotherapy, cancer immunosuppressive therapy, growth factors (except erythropoietin), radiation therapy (other than whole brain irradiation [WBI]) surgery or ablative therapy or investigational drugs/devices ≤28 days before first dose of trial treatment.
8. Subjects receiving high doses of corticosteroids must have been tapered to a stable dose at least 7 days before the first dose of trial treatment.
9. Tyrosine kinase inhibitor within 7 days prior to the first dose of trial treatment.
10. Subjects with overt leptomeningeal leukemia or central nervous system (CNS) lymphoma. Subjects must be free of CNS disease for a minimum of 2 months. Subjects with symptoms of CNS disease must have a negative diagnostic lumbar puncture prior to study enrollment.
11. Subjects with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
12. Baseline QTcF >480 ms. Note: This criterion does not apply to subjects with a left bundle branch block.
13. Subjects who have had a venous thromboembolic event requiring anticoagulation and who meet any of the following criteria:

    * Have been on a stable dose of anticoagulation for <1 month.
    * Have had a Grade 2, 3 or 4 hemorrhages in the last 30 days.
    * Are experiencing continued symptoms for their venous thromboembolic event.
14. Subjects with a history of liver disease as a result of alcohol abuse, chronic hepatitis, or other chronic liver disease (other than metastatic disease to the liver).
15. Subjects with positive HBsAg, HBcAb or HCV are excluded.
16. Subjects with a history of tuberculosis within the preceding two years.
17. Prior surgery affecting drug absorption or any gastrointestinal dysfunction that could alter drug absorption.
18. Subjects with a known hypersensitivity to bendamustine or rituximab.
19. Presence of active infection within 72 hours of treatment. Subjects with ongoing use of prophylactic antibiotics are eligible as long as there is no evidence of active infection and the antibiotic is not included on the list of prohibited medications.
20. Known diagnosis of human immunodeficiency virus (HIV).
21. Concurrent administration of medications or foods that are strong or moderate inhibitors or inducers of CYP3A.
22. Women who are pregnant or lactating.
23. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
24. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol or would impart excessive risk associated with study participation that would make it inappropriate for the subject to be enrolled.
25. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The number of adverse events, serious adverse events, and dose limiting toxicities as a measure of safety and tolerability | up to 12 months
  The maximum tolerated dose of IPI-145 defined as the optimal dose at which ≤1 of 6 patients experiences a DLT assessed by NCI CTCAE v4.0.

SECONDARY OUTCOMES:
Antitumor activity | Up to 5 years
  Preliminary information on antitumor activity of IPI-145 when combined with rituximab, or bendamustine/rituximab as measured by objective response rate, progression free survival and overall survival data

OTHER OUTCOMES:
PK of IPI-145 and its metabolites | Day 1
  Pharmacokinetics (PK) of IPI-145 and its metabolites when combined with rituximab or bendamustine/rituximab will be obtained by evaluating maximum concentration and area under the curve pre-dose and up to 6 hours post-dose.
PDx of IPI-145 | Up to 12 months
  Pharmacodynamics (PDx) of IPI-145 when combined with rituximab or bendamustine/rituximab will be evaluated by assessing chemokines and cytokines.
Molecular predictors of IPI-145 | Up to 12 months
  Develop molecular predictors of response when IPI-145 is combined with rituximab or bendamustine/rituximab by assessing protein expression and potential mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Flinn, M.D., Study Chair — SCRI
Locations (4):
- United States (4):
  - The Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Oklahoma University, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC, Nashville, Tennessee